CLINICAL TRIAL: NCT01462487
Title: Assessing the Safety of Inhaled Zanamivir Exposure in Pregnant Women
Brief Title: Safety of Inhaled Zanamivir in Pregnancy
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114791; WEUSRTP4948 (Other: GSK); EPI40649 (Other: GSK)
Record Dates: First submitted 2011-09-29; First posted 2011-10-31 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Influenza, Human
Keywords: Pregnancy safety; zanamivir; influenza
MeSH Terms: conditions — Influenza, Human | interventions — Therapeutics; Zanamivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pregnancy outcomes analysis group: Pregnant women evaluated for the following pregnancy outcomes: elective termination, spontaneous abortion (defined as spontaneous fetal loss at < 20 weeks' gestation), fetal death (defined as death of a fetus at > 20 weeks' gestation), premature birth (defined as a birth occurring at < 37 weeks' gestation), and live birth at term
  Interventions: Drug: Treatment with zanamivir
- Congenital anomalies analysis group: Infants evaluated for congenital anomalies
  Interventions: Drug: Treatment with zanamivir
- Treatment-emergent diagnoses analysis group: Pregnant women evaluated for treatment-emergent diagnoses
  Interventions: Drug: Treatment with zanamivir

INTERVENTIONS:
Drug: Treatment with zanamivir — Subjects treated with zanamivir

SUMMARY:
Zanamivir is a neuraminidase inhibitor that has demonstrated effectiveness against the pandemic H1N1 virus. Zanamivir was first authorized in Sweden in June 1999 and is approved in the European Union (EU) through mutual recognition. It is indicated for treatment and prevention of influenza in adults and children over the age of 5 years.

Zanamivir animal studies, conducted primarily in rabbits, showed a trend towards increased post-implantation loss, decreased fetal body weight, and increased minor fetal skeletal changes, although these effects were not statistically significant. Given the frequency, pattern and distribution of these effects, it was concluded that they were not related to zanamivir treatment. The summary of product characteristics for zanamivir states that it should not be used during pregnancy unless the potential benefit to the mother justifies the risk to the fetus.

Postmarketing data have shown no higher risk of malformation with oseltamivir than in the general population, but data on zanamivir are scarcer. Limited data are available on pregnancy outcomes with maternal exposure to zanamivir during pregnancy. From 01 August 2003 through 31 January 2009, 133 women were reported to have been treated with zanamivir while pregnant. Of these 133 pregnancies, 83 pregnancies were on-going or had been lost to follow-up (62.4%) at the time of the report; 43 resulted in a live birth with no apparent congenital anomalies (32.3%), 4 represented spontaneous abortions with no apparent congenital anomalies (3.0%), 2 were elective terminations with no apparent congenital anomalies (1.5%), and 1 was an ectopic pregnancy (<1%). The European Medicines Agency (EMA) has concluded that exposure to zanamivir during pregnancy does not represent a new safety risk to the fetus.

Published research has suggested that early antiviral treatment of pregnant H1N1 patients can improve outcomes. In a Center for Disease Control and Prevention (CDC) surveillance population of 788 pregnant influenza patients with disease onset between April and August 2009, the 384 with data on timing of antiviral treatment were observed to have significantly higher risk of adverse outcomes with later treatment ('intermediate', i.e. 3-4 days, n=84; 'late', i.e. > 4 days: n=81) than with early treatment (< 2 days: n=219). Compared with those given early treatment, those given intermediate treatment had almost 10 times the risk of death, and those given late treatment, more than 50 times. Intensive Care Unit (ICU) admission showed more than a 2-fold risk elevation with intermediate treatment and a six-fold elevation with late treatment, Respective elevations in risk of need for mechanical ventilation were almost 4-fold and more than 12-fold. The authors noted that the reason for treatment delays in this population are unknown, but could include reluctance on the part of clinicians and patients to expose the fetus to antiviral medications, as well as use of rapid influenza tests, which have shown low (10%-70%) sensitivity for H1N1.

As part of their ongoing epidemiologic safety monitoring initiatives requested by the EMA during the influenza pandemic of 2009-2010, GSK seeks to conduct a pregnancy safety study to better understand the safety of zanamivir in women exposed during pregnancy for either the treatment or prevention of influenza. This safety study will collect information from existing European databases with records of pregnant women exposed to these products and their pregnancy outcomes in order to assess the safety of these treatments in this population.

GSK is working with PPD as the contract research organization (CRO) to oversee conduct of this study, including data source management and payment, study design input, epidemiological advice, data transfer oversight and overall project management. The CRO will keep a record of all relevant personnel involved in the study. Additionally, PPD has a strategic alliance with World Health Information Science Consultants, LLC (WHISCON) (www.whiscon.com), an internationally recognized organization conducting post-approval drug safety and risk management epidemiology. WHISCON will be providing services related to protocol development as well as database-specific work plans, and will assist in analysis and interpretation of data.

The primary objective of this study is to evaluate the safety of zanamivir taken during pregnancy on 1) the outcome of the pregnancy, 2) congenital anomalies identifiable at or shortly after birth, and 3) treatment-emergent diagnoses in the mother occurring within 28 days of receipt of zanamivir.

The secondary objectives of this study are 1) to develop techniques for identifying influenza-like illness (ILI) in the participating data sources, and 2) to identify the characteristics of zanamivir recipients.

ELIGIBILITY:
Inclusion Criteria:

Pregnacy Outcomes and Treatment Emergent Diagnoses Analysis Groups:

* Pregnant women who have received treatment or prophylaxis regimens of zanamivir or have not received these products
* Pregnancy completion occurring from December 2009 through November 2010

Cogenital Anomalies Group:

* Live born infants of pregnant women included in the Pregnacy Outcomes and Treatment Emergent Diagnoses Analysis Groups

Exclusion Criteria:

* Women who received amantadine or rimantadine at any time during pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The observed population will include pregnant women who have received zanamivir and pregnant women who have not received influenza antiviral therapy.
  Subject pregnancies will be identified on the basis of pregnancy completion occurring from December 2009 through November 2010 and zanamivir exposure (or the absence of it). Follow-up data on live-born infants will be obtained at the time of delivery and for a maximum of 28 days after birth.
  The subject pregnancies' data will be obtained from the following four European data systems: Danish National Linked Databases, CSD MR UK (formerly known as EPIC), a subsidiary of Cegedim Strategic Data, PHARMO Network (Institute for Drug Outcomes Research), and Swedish Medical Birth Register.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcomes | Within 24 hours of birth
  Pregnancy outcomes including elective termination, spontaneous abortion (defined as spontaneous fetal loss at < 20 weeks' gestation), fetal death (defined as death of a fetus at > 20 weeks' gestation), premature birth (defined as a birth occurring at < 37 weeks' gestation), and live birth at term

SECONDARY OUTCOMES:
Congenital anomalies | Within 24 hours of birth
Treatment-emergent diagnoses in the mother | From the beginning of pregnancy through the end of pregnancy, an average of 9 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline